CLINICAL TRIAL: NCT04249284
Title: A Study to Evaluate the Pharmacokinetics of BMS-986165 Administered as Various Prototypic Solid Tablet Formulations in Healthy Subjects
Brief Title: Pharmacokinetics (Drug Levels in Blood) of BMS-986165 When Taken as Various Solid Tablet Prototypes by Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IM011-096
Record Dates: First submitted 2020-01-29; First posted 2020-01-30 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Healthy Participants
MeSH Terms: interventions — deucravacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment A : BMS-986165 (Experimental)
  Interventions: Drug: BMS-986165
- Treatment B: BMS-986165 prototype 1 (Experimental)
  Interventions: Drug: BMS-986165 prototype 1
- Treatment C: BMS-986165 prototype 2 (Experimental)
  Interventions: Drug: BMS-986165 prototype 2
- Treatment D: BMS-986165 prototype 2 (Experimental)
  Interventions: Drug: BMS-986165 prototype 2

INTERVENTIONS:
Drug: BMS-986165 — Specified dose on specified days
  Arms: Treatment A : BMS-986165
Drug: BMS-986165 prototype 1 — Specified dose on specified days
  Arms: Treatment B: BMS-986165 prototype 1
Drug: BMS-986165 prototype 2 — Specified dose on specified days
  Arms: Treatment C: BMS-986165 prototype 2; Treatment D: BMS-986165 prototype 2

SUMMARY:
The purpose of this study is to characterize the pharmacokinetics (the way the body absorbs, distributes and eliminates the drug) of BMS 986165 given in the form of various prototypes of solid tablets to healthy participants.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* In the opinion of the investigator, a healthy participant is determined by having no clinically significant deviation from normal in medical history, physical examination,electrocardiograms, vital signs, and clinical laboratory determinations.
* Body weight >= 50 kg at screening
* Women and men must agree to follow specific methods of contraception, if applicable

Exclusion Criteria:

* Any major surgery, per investigator's discretion, within 4 weeks of study drug administration
* Inability to tolerate oral medication
* History of allergy to BMS-986165 or related compounds

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) for BMS-986165 in plasma | Up to 18 days
Area under the plasma concentration-time curve from time 0 to the last quantifiable concentration (AUC(0-T)) for BMS-986165 in plasma | Up to 18 days
Area under the plasma concentration-time curve extrapolated to infinity (AUC(INF)) for BMS-986165 in plasma | Up to 18 days

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 23 days
Incidence of Serious Adverse Events (SAEs) | Up to 55 days
Number of clinically significant abnormalities in electrocardiogram (ECG) parameters | Up to 50 days
Number of participants with vital sign abnormalities in body temperature | Up to 50 days
Number of participants with vital sign abnormalities in respiratory rate | Up to 50 days
Number of participants with vital sign abnormalities in heart rate | Up to 50 days
Number of participants with vital sign abnormalities in blood pressure | Up to 50 days
Number of participants with clinical laboratory test abnormalities: Hematology tests | Up to 50 days
Number of participants with clinical laboratory test abnormalities: Clinical chemistry tests | Up to 50 days
Number of participants with clinical laboratory test abnormalities: Urinalysis tests | Up to 50 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Quotient Sciences Miami, Miami, Florida, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm